CLINICAL TRIAL: NCT03659123
Title: Prehabilitation & Rehabilitation in Oncogeriatrics: Adaptation to Deconditioning Risk and Accompaniment of Patients' With Cancer, a Multicenter Pilot Study
Brief Title: Prehabilitation & Rehabilitation in Oncogeriatrics: Adaptation to Deconditioning Risk and Accompaniment of Patients' With Cancer
Acronym: PROADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL16_0701
Record Dates: First submitted 2018-06-01; First posted 2018-09-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Old Injury
Keywords: Elderly; Prehabilitation; Cancer; Surgery
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention is designed to be implemented at different times of patients' care
  During the prehabilitation time:
  * Nutritional care
  * Total-body rehabilitation
  * Pharmaceutical conciliation During peri-operative time
  * Management of enhances rehabilitation of the elderly. During rehabilitation time
  * Nutritional, medication conciliation and functional follow-up During hospital-home transition time
  * Nutritional and functional follow-up
  * Optimisation of symptoms management: abdominal pain, nausea, vomiting…
  Interventions: Behavioral: standardized geriatric intervention

INTERVENTIONS:
Behavioral: standardized geriatric intervention — Nutritional care is based on:
  * A personalized evaluation of nutritional balance and nutritional needs of the patient
  * A weekly follow-up of weight and nutritional intake
  Total-body rehabilitation is based on:
  * 2 to 3 times a week: strength exercise
  * 2 to 3 times a week: endurance exercise, 20 to 45 min each sequence
  * 2 times a week: respiratory physiotherapy Pharmaceutical conciliation and optimization according STOPP/START criteria During peri-operative time, the nurse contacts the surgical team for transmission of patient's personal data, physical medication conciliation results During rehabilitation time and hospital-home transition time, the nurse contacts the rehabilitation team for transmission of patient's personal data and care course, physical (nutritional, functional and/or comorbidities), medication conciliation results.

SUMMARY:
With the conjunction of increased life expectancy and the increasing incidence of cancer with aging, older patient represent an increasing proportion of cancer patients. Increasing age is also associated with increased risk of co-morbidities as well as a decline of functional reserve of multiple organ systems, eventually leading in the context of the disease-and/or the treatment-related stress to functional deconditioning or organ failure.

Surgery or complex medico-surgical procedures - that associate chemotherapy and/or radiotherapy and surgery, can be considered as one proof-of principle of such risks, since major cancer surgery the older population is at higher risk of morbi-mortality and unplanned hospitalization for geriatric events In order to reduce complications after surgery, prehabilitation has often been considered, and 71% of the surgeons would accept a 4 weeks delay before surgery to improve patients' outcomes if shown to be beneficial. However, the actual level of evidence depends on the interventions: high for pre-operative nutrition, but low for physical exercise, due to heterogeneous programs with often bad adherence. In addition, geriatric validated interventions, in order to prevent iatrogenic event, may be added in a multi-interventional model of intervention.

DETAILED DESCRIPTION:
PROADAPT pilot study is a standardized geriatric intervention constructed on a multi-professional and multi-disciplinary basis after a systematic analysis of published data.

This intervention was designed to be implemented pragmatically in the centers according local habits in several distinct hospital contexts in different tumor contexts.

It consists in:

1. before surgery: a prehabilitation of the patients including a nutritional, physical and educational preparation;
2. during the hospitalization for surgery: an optimisation of their treatments through a pharmaceutical conciliation, educational interventions, standardization of surgical procedures and enhanced rehabilitation after surgery;
3. bridging and post-discharge interventions for hospital-to-home transition.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥70 year old OR patient ≥60 years with significant comorbid condition (modified Charlson index≥3) or disability (ADL score<6/6);
* Histologically or cytologically proven cancer.
* Life expectancy > 3 months.
* Written informed consent obtained
* Covered by a Health System where applicable.

Exclusion Criteria:

* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix or squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer.
* Patient unable to be regularly followed for any reason (geographic, familial, social, psychologic).
* Any mental or physical handicap at risk of interfering with the appropriate treatment.
* Any administrative or legal supervision where applicable

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Implementation of at least one item of PROADAPT standardized geriatric intervention of the program PROADAPT pilot study | 12 months
  Preoperative physical activity including strength and endurance exercise assessed by physical exercises accomplished under the supervision of a physiotherapist. Number of patients with at least 1 intervention achieved in the domain.
Implementation of at least one item of PROADAPT standardized geriatric intervention of the program PROADAPT pilot study | 12 months
  Nutrition guidelines before and after physical activity assessed by questionnaires. Number of patients with at least 1 intervention achieved in the domain.
Implementation of at least one item of PROADAPT standardized geriatric intervention of the program PROADAPT pilot study | 12 months
  Patient education and coaching assessed by questionnaires and visits. Number of patients with at least 1 intervention achieved in the domain
Implementation of at least one item of PROADAPT standardized geriatric intervention of the program PROADAPT pilot study | 12 months
  Achievement of standardized intervention procedures, according to the checklist established in consensus with surgeons. Number of patients with at least 1 intervention achieved in the domain
Implementation of at least one item of PROADAPT standardized geriatric intervention of the program PROADAPT pilot study | 12 months
  Rehabilitation assessed by questionnaires. Number of patients with at least 1 intervention achieved in the domain
Implementation of at least one item of PROADAPT standardized geriatric intervention of the program PROADAPT pilot study | 12 months
  Accomplishment of pharmaceutical medication conciliation and treatment optimization. Number of patients with at least 1 intervention achieved in the domain
Implementation of at least one item of PROADAPT standardized geriatric intervention of the program PROADAPT pilot study | 12 months
  Bridging interventions for hospital-to-home transition. Number of patients with at least 1 intervention achieved in the domain

SECONDARY OUTCOMES:
Post operative morbidity | 30 and 90 days
  Post operative morbidity according Clavien-Dindo classification
Post-operative morbidity | 90 days
  Post-operative morbidity according to NCI CTC v4.4
Therapeutic strategy | 12 months
  Treatment plan completion rate: Number of patients for whom the treatment plan was completed.
Progression-free Survival | 12 months
Post-treatment complication | 12 months
  Post-treatment complication grade≥3 according the National Cancer Institute Common Toxicity Criteria version 4 (NCI-CTC-v4)

CONTACTS AND LOCATIONS:
Overall Officials: Claire FALANDRY, MD, Principal Investigator — Hospices Civils de Lyon
Locations (10):
- France (10):
  - Centre Hospitalier de Chambéry, Chambéry
  - Centre hospitalier de Givors, Givors
  - Centre Hospitalier Edouard Herriot, Lyon
  - Hôpital Croix Rousse, Lyon
  - Centre hospitalier d'Annecy Genevois, Metz-Tessy
  - Centre Hospitalier Lyon Sud, Service d'Oncologie Médicale, Pierre-Bénite
  - Centre Hospitalier Lyon Sud, Service de Gériatrie, Pierre-Bénite
  - Centre hospitalier Universitaire de Saint Etienne, Saint-Etienne
  - Hôpital Nord-Ouest, Villefranche-sur-Saône
  - Clinique mutualiste Médipole, Villeurbanne

REFERENCES:
- [Result] Roche M, Ravot C, Malapert A, Paget-Bailly S, Garandeau C, Pitiot V, Tomatis M, Riche B, Galamand B, Granger M, Barbavara C, Bourgeois C, Genest E, Stefani L, Haine M, Castel-Kremer E, Morel-Soldner I, Collange V, Le Saux O, Dayde D, Falandry C; PROADAPT working group. Feasibility of a prehabilitation programme dedicated to older patients with cancer before complex medical-surgical procedures: the PROADAPT pilot study protocol. BMJ Open. 2021 Apr 2;11(4):e042960. doi: 10.1136/bmjopen-2020-042960. PMID 33811052